CLINICAL TRIAL: NCT04684940
Title: A Phase 1/2 Safety, Tolerability, and Efficacy Study of BMN 270, an Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A Patients With Active or Prior Inhibitors
Brief Title: Safety, Tolerability, and Efficacy Study of Valoctocogene Roxaparvovec in Hemophilia A With Active or Prior Inhibitors
Acronym: GENEr8-INH
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 270-205; 2019-003213-34 (EudraCT Number)
Record Dates: First submitted 2020-11-30; First posted 2020-12-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia A With Anti Factor VIII
Keywords: Gene Therapy; Clotting Disorders; Blood Disorder; Blood Coagulation Disorders; Inherited Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic DIseases; Factor VIII; Coagulants; Hemophilia A; AAV5 vector
MeSH Terms: conditions — Hemostatic Disorders; Hematologic Diseases; Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Hemophilia A | interventions — Valoctocogene Roxaparvovec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valoctocogene roxaparvovec Open Label (Experimental): Single administration of valoctocogene roxaparvovec at a dose of 6E13 vg/kg in Active Inhibitor Population (Part A) and Prior Inhibitor Population (Part B).
  Interventions: Biological: Valoctocogene roxaparvovec

INTERVENTIONS:
Biological: Valoctocogene roxaparvovec — Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A
  Other Names: BMN 270 (GENEr8)

SUMMARY:
This Phase I/II clinical study will evaluate the safety and efficacy of valoctocogene roxaparvovec in patients with severe haemophilia A and inhibitors to FVIII. Part A of the study will involve subjects who have active inhibitors to FVIII, and Part B involving subjects with a prior history of inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age with hemophilia A and documented prior residual FVIII activity ≤ 1 IU/dL including, but not limited to, at the time of detected inhibitors, at the time of signing the informed consent.
2. History of a positive inhibitor result with the first positive result at least 12 month prior to Screening.

   Part A: Demonstrated no immunological tolerance to exogenous FVIII. Part B: Demonstrated tolerance to exogenous FVIII and negative FVIII inhibitor screening titer < 0.6 BU.
3. Prophylactic or on-demand hemophilia therapy in the last 12 months. Bleeding, inhibitor & hemophilia therapy Hx over previous 12 months.
4. Sexually active participants must agree to use an acceptable method of effective contraception. Participants must agree to contraception use for at least 12 weeks post-infusion.
5. Willing to abstain from consumption of alcohol for at least the first 52 weeks following BMN 270 infusion.

Exclusion Criteria:

1. Detectable pre-existing antibodies to the AAV5 capsid.
2. Any evidence of active infection or any immunosuppressive disorder; patients with HIV infection and undetectable viral load are not excluded.
3. Currently undergoing, or plan to receive during the study, immune tolerance induction therapy or prophylaxis with FVIII (Part A only).
4. Significant renal dysfunction or liver dysfunction, infection or history of hepatic malignancy.
5. Evidence of any bleeding disorder not related to hemophilia A.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological males only
Enrollment: 10 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events, as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 after administration of BMN 270. | 60 months

SECONDARY OUTCOMES:
Change of the median Factor VIII activity. | 60 months
  Changes in the median Factor VIII activity (IU/mL) after administration of BMN 270 which will be measured using the chromogenic FVIII assay.
A change in Factor VIII inhibitor titer (Part A) after administration of BMN 270. | 60 months
  FVIII inhibitor titer will be measured using a chromogenic Nijmegen-Bethesda assay.
Absence of recurrence of Factor VIII inhibitors (Part B) after administration of BMN 270. | 60 months
  FVIII inhibitor titer will be measured using a chromogenic Nijmegen-Bethesda assay.
Change in the annualized utilization of hemophilia therapy after administration of BMN 270 | 60 months
Change in the annualized number of bleeding episodes requiring exogenous hemophilia therapy after administration of BMN 270. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — BioMarin Pharmaceutical
Locations (9):
- Children's Hospital Los Angeles, Los Angeles, California, United States
- Brazil (2):
  - Hemocentro Da UNICAMP, Campinas
  - Arthur De Siqueira Cavalcanti Hematology State Institute, Rio de Janeiro
- Chaim Sheba Medical Center, Ramat Gan, Israel
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea
- Taiwan (3):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Ege University School of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No